CLINICAL TRIAL: NCT05152654
Title: Is it Necessary to Fix Mesh in Laparoscopic Hernia Repair; Prospective Randomized Double-blinded Controlled Study
Brief Title: Is it Necessary to Fix Mesh in Laparoscopic Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Murat Baki YILDIRIM, assistant professor, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mesh fixation
Record Dates: First submitted 2021-09-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Inguinal Hernia; Pain, Acute; Pain, Chronic
MeSH Terms: conditions — Hernia, Inguinal; Acute Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Patients participating in the study will be divided into two groups. Patients with unilateral inguinal hernia will be determined according to the envelope selection method. Patients will not know which group are in. The patients in the first group will be fixed with 5 tackers while performing total extraperitoneal repair. While the patients in the second group are performing total extraperitoneal repair, no fixation will be made while placing the mesh.
Who Masked: Care Provider
Masking Description: Only the practicing surgeon will know which group the patients will be in until the end of the study. will not share this information with researchers and patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixation (No Intervention): Total extra peritoneal repair will be performed in this arm for the patients due to unilateral inguinal hernia. The 15x12 cm mesh will be marked with titanium clips from its 4 corners and placed in the hernia area. The mesh will be fixed to the hernia area by the non-absorbable tacker.This method is the method used routinely in the treatment of laparoscopic hernia today.
- Non-Fixation (Experimental): Total extra peritoneal repair will be performed in this arm for the patients due to unilateral inguinal hernia. The 15x12 cm mesh will be marked with titanium clips from its 4 corners and placed in the hernia area. The mesh will not be detected in any way.
  Interventions: Device: Tacker

INTERVENTIONS:
Device: Tacker — metallic staples used to fix the mesh
  Arms: Non-Fixation

SUMMARY:
Inguinal hernias are one of the most common diseases in general surgery practice. In a multicenter study conducted in Germany, inguinal hernia repair is one of the most common operations. Until the last 20 years, after Lichtenstein described tension-free mesh hernia repair, this method was the gold standard in inguinal hernia surgery. This method was advantageous in terms of both less recurrence and less postoperative pain compared to tension methods. With the development of minimally invasive surgery, laparoscopic hernia surgery was first described by Dr. Ger in 1992. Laparoscopic inguinal hernia repair is based on the principles of preperitoneal repair described by Stoppa in open surgery. Its advantages over laparoscopic surgery are; Less post-operative pain, rapid recovery, reduction in nerve damage and chronic pain, and reduced recurrence rate. However, the disadvantage is that the learning curve is longer and higher cost. Two commonly used laparoscopic inguinal hernia surgeries are Trans Abdominal Pre-Peritoneal (TAPP) and totally extraperitoneal (TEP) methods. Although both are preperitoneal repair methods, less intraperitoneal organ damage, less intra-abdominal adhesion formation, and no need for peritoneal sheath repair are the advantages of the TEP method. For this reason, TEP method has been the preferred method today. Various methods have been tried in order not to change the location of the mesh placed in the TEP method. Laparoscopic inguinal hernia is one of the most debated issues. The most common methods for fixation are tacker, tissue adhesive, or suturing the mesh. However, fixing the mesh using a tacker can cause chronic pain. Tissue adhesives are not preferred because tissue adhesives have high costs and sometimes cause allergic reactions. The method in which the mesh is sewn to the pubic bone is avoided by surgeons because it prolongs the operation time. To avoid chronic pain after surgery, the idea was not to fix the mesh. The major drawback of this method is that the mesh may slip and cause recurrence.This study aimed to reveal the difference between the amount of migration and the amount of post-operative pain between detecting the mesh and not detecting it

DETAILED DESCRIPTION:
The study will be conducted as a prospective, double-blind, randomized controlled study in the general surgery clinic of a university hospital. As a result of the power analysis calculated under Cohen's expert opinion, it was decided to include a total of 100 patients, 50 patients in order to reach 80% power with 0.50 effect size (medium effect) and 5% error (alpha=0.05). in each group. The study will continue by taking the consent of the patients and choosing from among the volunteer patients. The method by which the patients will be operated will be determined by choosing from a total of 100 (50 per group) sealed envelopes containing the group names. In the first (Fixation Group) group, inguinal hernia repair with the TEP method will be fixed with a mesh stapler. While inguinal hernia repair is performed with TEP method in the second (Non-Fixation Group) group, the mesh will not be fixed by any method. Exclusion criteria; It was determined as being younger than 18 years of age, having a comorbidity that prevented him from receiving general anesthesia, having had a previous lower abdominal surgery, having undergone previous inguinal hernia surgery, having bilateral inguinal hernia, scrotal hernia or strangulated hernia.

Creation of double blind; Patients will not be told which study group participants are in as a result of the envelope participants choose. In the postoperative follow-up of the patients, the researcher who recorded the parameters related to the study and provided the measurements will not know which group the patients are in.

Age, gender, comorbidity, smoking history and body mass index of the patients will be recorded on the preoperative forms. The surgery will be performed by a single surgeon according to the group chosen by the patients. The performing surgeon was a general surgeon with 5 years of active experience in laparoscopic hernia surgery and had performed both methods more than 200 times. Until the end of the study, only the surgeon will know which group the patients are in. The investigator evaluating the results of the study and the performing surgeon will not communicate about the study.

ELIGIBILITY:
Inclusion Criteria:

* being over 18 years old
* having a unilateral inguinal hernia

Exclusion Criteria:

* being under18 years old
* having comorbidity that prevents him from receiving general anesthesia
* having undergone previous lower abdominal surgery
* having previous surgery for inguinal hernia
* having bilateral inguinal hernia, scrotal hernia or strangulated hernia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
displacement of the mesh one day after surgery | one day after surgery
  It is the process of measuring how much the mesh placed in the surgery is displaced. Determining the distance of the titanium clips placed at the four corners of the mesh to the symphysis pubis and measuring the change in time intervals. Abdominal radiographs of the patients in both study arms will be taken one day after the operation, and the distance between the symphysis pubis and the titanium clips placed on the mesh will be recorded in millimeters.
displacement of the mesh one week after surgery | first week after surgery and 6th month after surgery
  It is the process of measuring how much the mesh placed in the surgery is displaced. Determining the distance of the titanium clips placed at the four corners of the mesh to the symphysis pubis and measuring the change in time intervals. Abdominal radiographs of the patients in both study arms will be taken one week after the operation, and the distance between the symphysis pubis and the titanium clips placed on the mesh will be recorded in millimeters.
displacement of the mesh six month after surgery | first week after surgery and 6th month after surgery
  It is the process of measuring how much the mesh placed in the surgery is displaced. Determining the distance of the titanium clips placed at the four corners of the mesh to the symphysis pubis and measuring the change in time intervals. Abdominal radiographs of the patients in both study arms will be taken 6 months after the operation, and the distance between the symphysis pubis and the titanium clips placed on the mesh will be recorded in millimeters.
Postoperative 24th hours pain | 24th hours after surgery
  Patients will be asked about their visual pain score at the postoperative 24th hour. In this scoring system, 0 represents the least pain and 10 represents the most pain. Visual Analogue Scale(VAS) :min 0 max:10 (0 is better)
Postoperative 6th months pain | 6th month after surgery
  Patients will be asked about their visual pain score at 6 months postoperatively. In this scoring system, 0 represents the least pain and 10 represents the most pain. Visual Analogue Scale(VAS) :min 0 max:10 (0 is better)

CONTACTS AND LOCATIONS:
Overall Officials: Murat B YILDIRIM, Principal Investigator — Hitit University
Locations (1):
- Hitit University, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Buyukasik K, Ari A, Akce B, Tatar C, Segmen O, Bektas H. Comparison of mesh fixation and non-fixation in laparoscopic totally extraperitoneal inguinal hernia repair. Hernia. 2017 Aug;21(4):543-548. doi: 10.1007/s10029-017-1590-2. Epub 2017 Feb 18. PMID 28214943
- [Result] Darwish A. A, Hegab A. A . Tack fixation versus nonfixation of mesh in laparoscopic transabdominal preperitonaeal hernia repair. Egyptian Journal of Surgery. 2016;35(4): 327-331. DOI: 10.4103/1110-1121.194729
- [Derived] Yildirim MB, Sahiner IT. The effect of mesh fixation on migration and postoperative pain in laparoscopic TEP repair: prospective randomized double-blinded controlled study. Hernia. 2023 Feb;27(1):63-70. doi: 10.1007/s10029-022-02587-w. Epub 2022 Mar 14. PMID 35286511